CLINICAL TRIAL: NCT03045198
Title: Effect of Azithromycin on Lipoproteins and Docosahexaenoic Acid in Patients With Cystic Fibrosis
Brief Title: Effect of Azithromycin on Fatty Acids in CF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Childrens' Hospital (Zentrum für Kinderheilkunde des Universitätsklinikum Bonn) (Other)
Collaborators: University of Bonn (Other); Goethe University (Other)
Responsible Party: Principal Investigator, Sabina Schmitt-Grohe, PD Dr Sabina Schmitt-Grohé, University Childrens' Hospital (Zentrum für Kinderheilkunde des Universitätsklinikum Bonn)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sylvia 253/12
Record Dates: First submitted 2017-02-02; First posted 2017-02-07 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: CF patients receive for 4 weeks Azithromycin. Study measures are assessed before and after 4 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Azithromycin (Experimental): oral Azithromycin 10 mg/kg Body weight, max. 500 mg every Monday, Wednesday and Friday for 4 weeks
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin
  Other Names: Zithromax

SUMMARY:
In collaboration with Dr.Birgit Alteheld, Institute of Nutrional Sciences of the university of Bonn, Germany the following effect is explored: Effect of a 4 week therapy with AZT on synthesis of lipoproteins as well as Docosahexaen and other fatty acids in patients with Cystic Fibrosis (CF). Moreover proinflammatory cytokines in blood and sputum are of interest.

DETAILED DESCRIPTION:
The macrolide azithromycin (AZT) is recommended by Flume in the CF pulmonary Guidelines for long-term treatment of patients with CF chronically colonized with Pseudomonas aeruginosa due to its immunomodulating properties . AZT causes a significant reduction of the proinflammatory cytokine Lipopolysaccharid binding protein (LBP) according to Steinkamp and Schmitt-Grohé. There is an inverse correlation between LBP and lung function. Moreover Schmitt-Grohé and coworkers provided evidence of a positive correlation between the lipoprotein HDL and lung function. Ribeiro and coworkers found an increased expression of Lipid/Cholesterol genes of primary human airway epithelial cultures after treatment with AZT. Freedman and coworkers were able to show decreased levels of Docosahexaen acid in CF patients.

The aim of this study is to explore the impact of a 4 week trial of AZT on lipoprotein and fatty acids (docosahexaen acid etc.) synthesis.

Delta F508 homozygous patients receive AZT (10 mg/kg body weight resp. max 500 mg) every Monday, Wednesday and Friday for 4 weeks. 20 patients (age 10-60 years) will be recruited. Fatty acids (blood), cytokines (whole blood and induced sputum) and clinical parameters are assessed before and 4 weeks after AZT treatment.

ELIGIBILITY:
Inclusion Criteria:

* Delta 508 homozygous and regularly visiting the CF outpatient clinic Bonn

Exclusion Criteria:

* clinical or laboratory signs (CRP > 20 mg/L) of an exacerbation,
* treatment with systemic steroids 14 days preceeding this trial
* elevated liver function tests (> twice normal range)

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-03; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Lipoproteins in Serum (after overnight fast) | Day 0 (before azithromycin), Day 28 (day 28 of azithromycin treatment)
  VLDL,LDL,HDL, Cholesterin
Fatty acids in EDTA-Plasma and erythrocyte membranes (after overnight fast) | Day 0 (before azithromycin), Day 28 (day 28 of azithromycin treatment)
  linol acid, arachidon acid, Alpha linolen acid, eicosapentaen acid, Docoshexaen acidsdocosahexaen acid

SECONDARY OUTCOMES:
Cytokines in induced sputum and whole blood | Day 0 (before azithromycin), Day 28 (day 28 of azithromycin treatment)
  Lipopolysaccharid binding Protein (LBP), interleukin-8 (IL-8) und Tumor necrosis factor Alpha (TNF Alpha)
ICAM1 (Serum) | Day 0 (before azithromycin), Day 28 (day 28 of azithromycin treatment)
Matrixmetalloprotease 9 (Serum) | Day 0 (before azithromycin), Day 28 (day 28 of azithromycin treatment)
WBC + CRP, IgE, RAST Aspergillus fum, ECP (Serum), Carotin, Vitamin E | Day 0 (before azithromycin), Day 28 (day 28 of azithromycin treatment)
Shwachman-Score | Day 0
  Clinical score
Body weight, length | Day 0 (before azithromycin), Day 28 (day 28 of azithromycin treatment)
Lung function test | Day 0 (before azithromycin), Day 28 (day 28 of azithromycin treatment)
  VC, FEV1, MEF 25
Nutrition protocol | For 7 days before day 0 and day 28
  Evaluation of Food intake and calculation of fat composition, Protein etc.
Resolvins in EDTA plasma | Day 0 (before azithromycin), Day 28 (day 28 of azithromycin treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Schmitt-Grohé, MD, Principal Investigator — University Children's Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Freedman SD, Blanco PG, Zaman MM, Shea JC, Ollero M, Hopper IK, Weed DA, Gelrud A, Regan MM, Laposata M, Alvarez JG, O'Sullivan BP. Association of cystic fibrosis with abnormalities in fatty acid metabolism. N Engl J Med. 2004 Feb 5;350(6):560-9. doi: 10.1056/NEJMoa021218. PMID 14762183
- [Background] Steinkamp G, Schmitt-Grohe S, Doring G, Staab D, Pfrunder D, Beck G, Schubert R, Zielen S. Once-weekly azithromycin in cystic fibrosis with chronic Pseudomonas aeruginosa infection. Respir Med. 2008 Nov;102(11):1643-53. doi: 10.1016/j.rmed.2008.03.009. Epub 2008 Aug 12. PMID 18701270
- [Background] Schmitt-Grohe S, Hippe V, Igel M, von Bergmann K, Posselt HG, Krahl A, Smaczny C, Wagner TO, Nikolazik W, Schubert R, Lentze MJ, Zielen S. Lipopolysaccharide binding protein, cytokine production in whole blood, and lipoproteins in cystic fibrosis. Pediatr Res. 2005 Nov;58(5):903-7. doi: 10.1203/01.PDR.0000182598.98167.24. Epub 2005 Sep 23. PMID 16183806
- [Background] Flume PA, O'Sullivan BP, Robinson KA, Goss CH, Mogayzel PJ Jr, Willey-Courand DB, Bujan J, Finder J, Lester M, Quittell L, Rosenblatt R, Vender RL, Hazle L, Sabadosa K, Marshall B; Cystic Fibrosis Foundation, Pulmonary Therapies Committee. Cystic fibrosis pulmonary guidelines: chronic medications for maintenance of lung health. Am J Respir Crit Care Med. 2007 Nov 15;176(10):957-69. doi: 10.1164/rccm.200705-664OC. Epub 2007 Aug 29. PMID 17761616
- [Background] Ribeiro CM, Hurd H, Wu Y, Martino ME, Jones L, Brighton B, Boucher RC, O'Neal WK. Azithromycin treatment alters gene expression in inflammatory, lipid metabolism, and cell cycle pathways in well-differentiated human airway epithelia. PLoS One. 2009 Jun 5;4(6):e5806. doi: 10.1371/journal.pone.0005806. PMID 19503797